CLINICAL TRIAL: NCT00967707
Title: Population Pharmacokinetic and Pharmacodynamic Modeling of Gabapentin in Neuropathic Pain - Effect of Adjuvant Pharmacotherapy
Brief Title: Population Pharmacokinetic-pharmacodynamic (PK-PD) Modeling of Co-administered Gabapentin in Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBPPKPD-09; EudraCT number 2009-010783-41
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-09

CONDITIONS: Post-traumatic Neuropathic Pain
MeSH Terms: interventions — Gabapentin; Venlafaxine Hydrochloride; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin + venlafaxine (Active Comparator)
  Interventions: Drug: gabapentin and venlafaxine
- Gabapentin + donepezil (Active Comparator)
  Interventions: Drug: gabapentin and donepezil

INTERVENTIONS:
Drug: gabapentin and venlafaxine — Week 1-6: Gabapentin monotherapy (titration to individual maximum tolerated dose or maximum 800 mg 3 times daily).
  Week 7-12: Venlafaxine 75 mg once daily is added.
  Arms: Gabapentin + venlafaxine
Drug: gabapentin and donepezil — Week 1-6: Gabapentin monotherapy (titration to individual maximum tolerated dose or maximum 800 mg 3 times daily).
  Week 7-12: Donepezil 5 mg once daily is added.
  Arms: Gabapentin + donepezil

SUMMARY:
The primary objective of this study is to develop a pharmacokinetic (PK) and a pharmacokinetic-pharmacodynamic (PK-PD) model for gabapentin in patients with neuropathic pain.

The secondary objectives are to investigate whether adjuvant therapy of venlafaxine or donepezil contributes to 1) improved analgesic efficacy and 2) improved health-related quality of life (assessed by the SF-36 questionnaire) in neuropathic pain patients treated with gabapentin.

DETAILED DESCRIPTION:
Neuropathic pain is estimated to affect 2-3 % of the population and the condition is difficult to treat with conventional analgesics. The drug of first choice is typically a tricyclic antidepressant drug (TCA) or the antiepileptic drug gabapentin. TCAs have well-documented effects, but the use is commonly interrupted due to intolerable adverse effects. Gabapentin, on the other hand, is generally well tolerated in patients. Clinical trials have proven that gabapentin is efficacious for neuropathic pain of various origins. Nevertheless, monotherapy is seldom sufficient for the management of severe neuropathic pain. Combination therapy, e.g. of gabapentin and an analgesic with complementary mechanism of action, may be a rational strategy to obtain improved results at lower doses and with fewer side effects. Although many neuropathic pain patients receive a combination of drugs, there is an absence of clinical evidence for optimal drug combinations.

Gabapentin binds to the alpha-2-delta subunit on presynaptic voltage-gated calcium channels, which results in modulation of the release of neurotransmitters from presynaptic nerve terminals. Recent studies in animal models of neuropathic pain have shown that gabapentin is effective on supraspinal structures, to activate the descending pain inhibitory noradrenergic-cholinergic cascade. Thus, it might be possible to potentiate the analgesic effect of gabapentin by concomitant administration of a drug able to prolong the action of noradrenaline or acetylcholine in the synapse cleft. In this study, the adjuvant effect of the noradrenaline and serotonin reuptake inhibitor venlafaxine and the cholinesterase inhibitor donepezil will be investigated in neuropathic pain patients treated with gabapentin.

The study consists of two periods. All patients are treated with gabapentin in the first period, and receive randomised adjuvant therapy of venlafaxine or donepezil in the second period. Repeated pain intensity ratings and blood samples for analysis of gabapentin plasma concentrations will be collected over one dosing interval of gabapentin at the end of each period.

Data will be analysed by means of nonlinear mixed effect modeling. The NONMEM programme will be used to develop models describing the PK and the PK-PD relationship of gabapentin in patients with neuropathic pain. The potential effect of concomitant treatment with venlafaxine or donepezil will be evaluated by covariate analysis in the developed PK and PK-PD models of gabapentin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-traumatic neuropathic pain
* Spontaneous pain intensity ≥ 40 on VAS or ≥ 4 on NRS
* Man or woman ≥ 18 years old
* Informed consent to study participation

Exclusion Criteria:

* Presence of other type of pain as strong as or stronger than the neuropathic pain
* Impaired kidney function (GFR < 30 ml/min)
* Uncontrolled cardiovascular disease/hypertonia
* Uncontrolled narrow-angle glaucoma
* Uncontrolled pulmonary disease
* Epilepsia
* Pregnancy
* Nursing
* Woman of childbearing potential not using contraception or planning to become pregnant during the study period
* Disability to understand and cooperate with study procedures
* Allergy to study medications
* Concomitant participation in other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity scorings on Numerical Rating Scale (NRS). Plasma concentrations of gabapentin. | 0 - 8 hours follwing dose intake of gabapentin. during steady state

SECONDARY OUTCOMES:
Health-related quality of life assessed by SF-36. Pain according to McGill Pain Questionnaire. | Minimum 6 weeks following initiation of gabapentin and combination therapy, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Butler, MD, Principal Investigator — Uppsala University
Locations (1):
- Multidisciplinary Pain Centre, Uppsala University Hospital, Uppsala, Sweden